CLINICAL TRIAL: NCT05999916
Title: A Prospective, Single-Arm, Monocentric Pilot Study to Evaluate the Safety and Feasibility of Transcranial Alternate Current Stimulation With the Miamind Neurostimulator in Healthy Participants
Brief Title: Evaluate the Safety and Feasibility of tACS With the Miamind Neurostimulator in Healthy Participants
Acronym: MindStim
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bottneuro AG (Industry)
Collaborators: Hemex AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: BTN-100
Record Dates: First submitted 2023-08-03; First posted 2023-08-21 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Healthy Participants; Healthy Population
Keywords: Alzheimer Disease; tACS; Memory Problems; Cognitive Impairment; Cognitive Performance; Safety and Tolerability; Feasibility
MeSH Terms: conditions — Alzheimer Disease; Memory Disorders; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: The present study aims to assess the safety and feasibility of employing repeated (4 sessions at 4 days) transcranial alternating current stimulation (tACS) through the utilization of the Miamind Neurostimulator in a cohort of healthy participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 60 min session of 40Hz tACS by Miamind Neurostimulator (Experimental): The clinical study will enroll eight (8) participants who will undergo four (4) tACS sessions (one per day) within 4 consecutive days. The tACS intervention will last 60 min in total. The stimulation frequency will be 40 Hz with max 1 mA/electrode and total of max 2 mA across all active electrodes (peak-to-baseline).
  Interventions: Device: Personalized Miamind Neurostimulator

INTERVENTIONS:
Device: Personalized Miamind Neurostimulator — 60 min. 40 Hz max. 1mA / electrode & total of max. 2 mA across all electrodes. 30- s ramp-up personalised intervention based on individual modelling of electric field distribution to maximise therapeutic effect in the target region. Three target regions, consecutively stimulated (20min each).

SUMMARY:
The present study aims to assess the safety and feasibility of repeated transcranial alternating current stimulation (tACS) by the Miamind Neurostimulator in a cohort of healthy participants. Based on the findings of this investigation, subsequent clinical trials assessing the efficiency of tACS by the Miamind Neurostimulator for treatment of Alzheimer's Disease will be conducted.

DETAILED DESCRIPTION:
The pathological hallmarks of Alzheimer's Disease (AD) are extracellular amyloid-β (Aβ) plaques and intracellular neurofibrillary tangles of hyperphosphorylated tau deposition in the brain together with neuroinflammation and microglial activation. These alterations lead to synaptic dysfunction, neuronal loss, and subsequently to brain circuit and brain oscillation disruption, resulting in cognitive decline. Recent studies have shown a positive effect of neural entrainment at gamma frequency (30-80 Hz). Transcranial alternating current stimulation (tACS) utilizes low amplitude alternating currents, allowing for frequency and region-specific brain oscillation entrainment showing positive results regarding improvement of cognitive functions in healthy participants and Alzheimer's Disease patients. Miamind Neurostimulator is a patient specific MRI-based 3D printed medical device that permits electrical stimulation and recording on up to 32 electrode channels and thus allows for simultaneous, multifocal, and targeted brain stimulation. tACS is non- invasive, well tolerated by users and considered safe with no persistent adverse events reported.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who are overtly healthy as determined by medical evaluation including medical history and physical examination.
2. Able and willing to provide voluntary written Informed Consent and sign the ICF to participate in the study prior to any study-related procedure.
3. Must have the ability to comply with protocol-related tests, appointments, and procedures.
4. Age over 18 years old.
5. Knowledge of the German language (B1 or higher).
6. No history of intellectual or learning disability; at least 8 grades of school.
7. Non-disturbing hairstyle or headdress that enables electrode contact with the scalp judged by the investigator.

Exclusion Criteria:

1. Any acute or chronic disease/disorder (e.g., cerebral, psychiatric, cardiovascular, pulmonary, metabolic, skin etc.)
2. History of traumatic brain injury or other diseases of the central nervous system.
3. History of seizures, diagnosis of epilepsy, or abnormal (epileptiform) EEG, or immediate (1st-degree relative) family history of epilepsy.
4. Diagnosis of substance abuse.
5. Participant is under the influence of alcohol, and consumption of narcotics or benzodiazepines, or other sleeping medications prior to the procedure.
6. All female participants that are not post-menopausal (defined as at least 12 months of spontaneous amenorrhea in women over 45 years old) or surgically sterile (e.g. bilateral tubal ligation, hysterectomy, bilateral oophorectomy) will be required to have a pregnancy test; any participant who is pregnant or breastfeeding will not be enrolled in the study.
7. Metal implants (excluding dental fillings) or devices such as a pacemaker, cardioverter defibrillator, medication pump, nerve stimulator, Transcutaneous Electrical Nerve Stimulator (TENS) unit, ventriculoperitoneal shunt, and cochlear implant, unless cleared by the study MD.
8. Contraindications for undergoing MRI.
9. Ongoing participation in any other interventional clinical study with an investigational drug or another MD within the 30 days preceding and during the present investigation.
10. Participants not suitable for the study based on a holistic consideration of the participant's history and the PI's medical expertise.

No vulnerable subject is enrolled on this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-12-27 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-03-22 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of Treatment-Emergent Adverse Events | up to 2 weeks
  Safety of the Treatment defined as the proportion of study participants free of serious adverse device effects and unanticipated serious adverse device effects (SADE and USADE) assessed via a safety questionnaire and medical evaluation.

SECONDARY OUTCOMES:
Safety and comfort: questionnaire | up to 2 weeks
  Adverse Events and comfort of tACS and the medical device are reported by questionnaires following stimulation of each target region at visit °3 & °4 and following sequential stimulation of multiple target regions at visit °5 & °6.
Evaluation of functional impact of tACS on Attention and Concentration: d2-R attention test | up to 2 weeks
  Changes in d2-R attention test are reported to document the functional impact of tACS on concentration and attention before and after stimulation of each target region at visit °3 & °4 and before and after sequential stimulation of multiple target regions at visit °5 & °6.
  The d2-R attention test measures processing speed, rule compliance, and quality of performance as estimation of attention and concentration and scores them as the following separate items: speed, concentration, carefulness. Each item is scored from 20-80. A higher score indicates better performance.
Evaluation of functional impact of tACS on oscillatory activity: Electroencephalography (EEG) | up to 2 weeks
  Quantification of EEG measurements to document the functional impact of tACS on oscillatory activity in individual frequency bands (delta, theta, alpha, beta, gamma) and EEG-biomarkers (alpha peak frequency, Vigilance) before and after stimulation of each target region at visit °3 & °4 & °5 & °6.
Cognitive Evaluation: Montreal Cognitive Assessment (MoCA) | up to 2 weeks
  MoCA scores are documented before and after visit °3 and after visit °6 to evaluate the impact of repeated tACS on cognitive performance.
  The MoCA has a total scoring range of 0-30, with the score based on the number of correct answers made in each of the 7 following items: Visuospatial/Executive, Naming, Memory/delayed recall, Attention, Language, Abstraction, Orientation. Sub-scores and total score are reported.
  A lower total score indicate greater cognitive impairment.
Participant coherence and satisfaction questionnaire | up to 2 weeks
  The subjective impression and satisfaction of the participant regarding the device and the intervention is documented using a one-time questionnaire at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Alois Hopf, PhD, Study Chair — Bottneuro AG
Locations (1):
- Universitätsspital Basel, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Background] Antal A, Alekseichuk I, Bikson M, Brockmoller J, Brunoni AR, Chen R, Cohen LG, Dowthwaite G, Ellrich J, Floel A, Fregni F, George MS, Hamilton R, Haueisen J, Herrmann CS, Hummel FC, Lefaucheur JP, Liebetanz D, Loo CK, McCaig CD, Miniussi C, Miranda PC, Moliadze V, Nitsche MA, Nowak R, Padberg F, Pascual-Leone A, Poppendieck W, Priori A, Rossi S, Rossini PM, Rothwell J, Rueger MA, Ruffini G, Schellhorn K, Siebner HR, Ugawa Y, Wexler A, Ziemann U, Hallett M, Paulus W. Low intensity transcranial electric stimulation: Safety, ethical, legal regulatory and application guidelines. Clin Neurophysiol. 2017 Sep;128(9):1774-1809. doi: 10.1016/j.clinph.2017.06.001. Epub 2017 Jun 19. PMID 28709880
- [Background] Nissim NR, McAfee DC, Edwards S, Prato A, Lin JX, Lu Z, Coslett HB, Hamilton RH. Efficacy of Transcranial Alternating Current Stimulation in the Enhancement of Working Memory Performance in Healthy Adults: A Systematic Meta-Analysis. Neuromodulation. 2023 Jun;26(4):728-737. doi: 10.1016/j.neurom.2022.12.014. Epub 2023 Feb 8. PMID 36759231
- [Background] Menardi A, Rossi S, Koch G, Hampel H, Vergallo A, Nitsche MA, Stern Y, Borroni B, Cappa SF, Cotelli M, Ruffini G, El-Fakhri G, Rossini PM, Dickerson B, Antal A, Babiloni C, Lefaucheur JP, Dubois B, Deco G, Ziemann U, Pascual-Leone A, Santarnecchi E. Toward noninvasive brain stimulation 2.0 in Alzheimer's disease. Ageing Res Rev. 2022 Mar;75:101555. doi: 10.1016/j.arr.2021.101555. Epub 2021 Dec 30. PMID 34973457
- [Background] Benussi A, Cantoni V, Grassi M, Brechet L, Michel CM, Datta A, Thomas C, Gazzina S, Cotelli MS, Bianchi M, Premi E, Gadola Y, Cotelli M, Pengo M, Perrone F, Scolaro M, Archetti S, Solje E, Padovani A, Pascual-Leone A, Borroni B. Increasing Brain Gamma Activity Improves Episodic Memory and Restores Cholinergic Dysfunction in Alzheimer's Disease. Ann Neurol. 2022 Aug;92(2):322-334. doi: 10.1002/ana.26411. Epub 2022 Jun 6. PMID 35607946
- [Background] Dhaynaut M, Sprugnoli G, Cappon D, Macone J, Sanchez JS, Normandin MD, Guehl NJ, Koch G, Paciorek R, Connor A, Press D, Johnson K, Pascual-Leone A, El Fakhri G, Santarnecchi E. Impact of 40 Hz Transcranial Alternating Current Stimulation on Cerebral Tau Burden in Patients with Alzheimer's Disease: A Case Series. J Alzheimers Dis. 2022;85(4):1667-1676. doi: 10.3233/JAD-215072. PMID 34958021
- [Background] Sprugnoli G, Munsch F, Cappon D, Paciorek R, Macone J, Connor A, El Fakhri G, Salvador R, Ruffini G, Donohoe K, Shafi MM, Press D, Alsop DC, Pascual Leone A, Santarnecchi E. Impact of multisession 40Hz tACS on hippocampal perfusion in patients with Alzheimer's disease. Alzheimers Res Ther. 2021 Dec 20;13(1):203. doi: 10.1186/s13195-021-00922-4. PMID 34930421
- [Derived] Joodaki M, Rodgers G, Hopf A, Koller MR, Guzman R, Santarnecchi E, Vogerl JS, Ferchow J, Ruffner A, Funken M, Meboldt M, Osmani B. A patient-specific, 3D printed neurostimulator enabling focal transcranial electrical stimulation and EEG at home. J Neuroeng Rehabil. 2025 Nov 24;22(1):248. doi: 10.1186/s12984-025-01769-8. PMID 41287086
- See also: Bottneuro Website — http://bottneuro.ch/en